CLINICAL TRIAL: NCT03745287
Title: A Phase 1/2/3 Study to Evaluate the Safety and Efficacy of a Single Dose of Autologous CRISPR-Cas9 Modified CD34+ Human Hematopoietic Stem and Progenitor Cells (CTX001) in Subjects With Severe Sickle Cell Disease
Brief Title: A Safety and Efficacy Study Evaluating CTX001 in Subjects With Severe Sickle Cell Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: CRISPR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTX001-121
Record Dates: First submitted 2018-11-09; First posted 2018-11-19 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease; Hematological Diseases; Hemoglobinopathies
MeSH Terms: conditions — Anemia, Sickle Cell; Hematologic Diseases; Hemoglobinopathies | interventions — exagamglogene autotemcel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX001 (Experimental): CTX001 (autologous CD34+ hHSPCs modified with CRISPR-Cas9 at the erythroid lineage-specific enhancer of the BCL11A gene). Subjects will receive a single infusion of CTX001 through a central venous catheter.
  Interventions: Biological: CTX001

INTERVENTIONS:
Biological: CTX001 — Administered by IV infusion following myeloablative conditioning with busulfan.
  Other Names: Exagamglogene autotemcel; Exa-cel

SUMMARY:
This is a single-arm, open-label, multi-site, single-dose Phase 1/2/3 study in subjects with severe sickle cell disease (SCD). The study will evaluate the safety and efficacy of autologous CRISPR-Cas9 Modified CD34+ Human Hematopoietic Stem and Progenitor Cells (hHSPCs) using CTX001.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of severe sickle cell disease as defined by:
* Documented severe sickle cell disease genotype
* History of at least two severe vaso-occlusive crisis events per year for the previous two years prior to enrollment
* Eligible for autologous stem cell transplant as per investigators judgment

Key Exclusion Criteria:

* An available 10/10 human leukocyte antigen (HLA)-matched related donor
* Prior hematopoietic stem cell transplant (HSCT)
* Clinically significant and active bacterial, viral, fungal, or parasitic infection

Other protocol defined inclusion/exclusion criteria may apply

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have not experienced any severe vaso-occlusive crisis (VOC) for at least 12 consecutive months (VF12) | From 60 days after last RBC transfusion up to 2 years after CTX001 infusion
Proportion of subjects with engraftment (first day of three consecutive measurements of absolute neutrophil count [ANC] ≥500/µL on three different days) | Within 42 days after CTX001 infusion
Time to engraftment | From CTX001 infusion up to 2 years after CTX001 infusion
Frequency and severity of collected adverse events (AEs) | From screening to 2 years after CTX001 infusion
Incidence of transplant-related mortality (TRM) within 100 days after CTX001 infusion | Within 100 days after CTX001 infusion
Incidence of TRM within 1 year after CTX001 infusion | Within 1 year after CTX001 infusion
All-cause mortality | 2 years after mobilization

SECONDARY OUTCOMES:
Proportion of subjects free from inpatient hospitalization for severe VOCs sustained for at least 12 months (HF12) | From 60 days after last RBC transfusion up to 2 years after CTX001 infusion
Proportion of subjects who have not experienced any severe VOC for at least 9 consecutive months (VF9) any time after CTX001 infusion | From 60 days after last RBC transfusion up to 2 years after CTX001 infusion
Proportion of subjects with 90 percent (%), 80%, 75% or 50% reduction in annualized rate of severe VOCs | From 60 days after last RBC transfusion up to 2 years after CTX001 infusion
Relative change from baseline in annualized rate of severe VOCs | From 60 days after last RBC transfusion up to 2 years after CTX001 infusion
Duration of severe VOC free in subjects who have achieved VF12 | From 60 days after last RBC transfusion up to 2 years after CTX001 infusion
Relative Change from baseline in rate of inpatient hospitalization for severe VOCs | From 60 days after last RBC transfusion up to 2 years after CTX001 infusion
Relative change from baseline in annualized duration of hospitalization for severe VOCs | From 60 days after last RBC transfusion up to 2 years after CTX001 infusion
Proportion of subjects with sustained HbF ≥20% for at least 3 months | From 60 days after last RBC transfusion up to 2 years after CTX001 infusion
Proportion of subjects with sustained HbF ≥20% for at least 12 months | From 60 days after last RBC transfusion up to 2 years after CTX001 infusion
Proportion of subjects with sustained HbF ≥20% for at least 6 months | From 60 days after last RBC transfusion up to 2 years after CTX001 infusion
Change in number of units of RBC transfused for SCD-related indications | 6 months up to 2 years after CTX001 infusion
HbF concentration over time | 1 month up to 2 years after CTX001 infusion
Hb concentration over time | From the time of CTX001 up to 2 years after CTX001 infusion
Change from baseline in indirect bilirubin over time | From baseline (pre-infusion) up to 2 years after CTX001 infusion
Change from baseline in reticulocyte count over time | From baseline (pre-infusion) up to 2 years after CTX001 infusion
Change from baseline in haptoglobin over time | From baseline (pre-infusion) up to 2 years after CTX001 infusion
Change from baseline in lactate dehydrogenase over time | From baseline (pre-infusion) up to 2 years after CTX001 infusion
Proportion of alleles with intended genetic modification present in peripheral blood leukocytes over time | 1 month up to 2 years after CTX001 infusion
Proportion of alleles with intended genetic modification present in CD34+ cells of bone marrow over time | 6 months up to 2 years after CTX001 infusion
Change in patient-reported outcome (PRO) over time assessed using weekly pain-scale (11-point numerical rating scale [NRS]) | 3 months up to 2 years after CTX001 infusion
  The NRS is a 1-dimensional measure of reporting intensity of pain. The score of NRS ranges from 0 to 10 points, with higher values indicating a higher level of pain.
Change in PRO over time assessed using EuroQol quality of life scale (EQ-5D-5L) | 3 months up to 2 years after CTX001 infusion
  The EQ-5D-5L Questionnaire consists of the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The EQ-5D comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and 5 levels: no problems to extreme problems. The subject marks the most appropriate statement in each dimension, resulting in a 1-digit number for that dimension. The digits can be combined in a 5-digit number describing the subject's health state. The EQ VAS records the subject's self-rated health on a 100-point VAS, endpoints labelled "the best health you can imagine" and "the worst health you can imagine"
Change in PRO over time assessed using EQ-5D-Youth (EQ-5D-Y) | 3 months up to 2 years after CTX001 infusion
Change in PRO over time assessed using functional assessment of cancer therapy-bone marrow transplant (FACT-BMT) questionnaire | 3 months up to 2 years after CTX001 infusion
  The FACT-BMT Questionnaire includes physical, social, family, emotional, and functional well-being, and treatment specific concerns of bone marrow transplantation. Each statement has a 5-point Likert-type response scale ranging from 0=not at all to 4=very much. The subject marks one number per line as it applies to the past 7 days. Questionnaires are then scored; the higher the score, the better the quality of life.
Change in PRO over time assessed using adult sickle cell quality of life measurement system (ASCQ-Me) | 3 months up to 2 years after CTX001 infusion
  ASCQ-Me comprises measures to assess physical, mental and social health along with information on severity of disease. It includes the following domains: emotional impact, pain impact, pain episodes, sleep impact, social functioning impact, stiffness impact and SCD medical history checklist. ASCQ-Me domains are scored using T-score metric with mean of 50 for reference population and SD of 10. Higher scores indicate healthier status.
Change in PRO over time assessed using pediatric quality of life inventory (PedsQL) | 3 months up to 2 years after CTX001 infusion
Change in PRO over time assessed using PedsQL sickle cell disease module | 3 months up to 2 years after CTX001 infusion

CONTACTS AND LOCATIONS:
Locations (17):
- United States (9):
  - Lucile Packard Children's Hospital of Stanford University, Palo Alto, California
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Illinois at Chicago Hospitals and Health Systems, Chicago, Illinois
  - Columbia University Medical Center (21+ years), New York, New York
  - Columbia University Medical Center (≤21 years), New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial Medical Center/ Sarah Cannon Center for Blood Cancers, Nashville, Tennessee
  - Methodist Children's Hospital/Texas Transplant Institute, San Antonio, Texas
- Hopital Universitaire des Enfants Reine Fabiola (HUDERF), Brussels, Belgium
- The Hospital for Sick Children, Toronto, Canada
- Hopital Necker Enfants Malades, Paris, France
- Germany (2):
  - University Hospital Duesseldorf, Düsseldorf
  - Regensburg University Hospital, Clinic and Polyclinic for Paediatric and Adolescent Medicine, Paediatric Haemotology, Oncology and Stem Cell Transplantation, Regensburg
- Dipartimento di Onco-Ematologia e Terapia Cellulare e Genica Ospedale Pediatrico Bambino Gesu - IRCCS, Rome, Italy
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London
  - Royal London and St Bartholomew's Hospital, Pathology and Pharmacy Building, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma A, Locatelli F, Bhatia M, Molinari L, Mapara MY, Liem RI, Dedeken L, Wall D, Eckrich MJ, Kuo KHM, Smith W, Imren S, Kohli P, Li N, Liu T, Rubin J, Hobbs W, Grupp SA, Frangoul H. Improvements in health-related quality of life in patients with severe sickle cell disease after exagamglogene autotemcel. Blood Adv. 2025 Dec 23;9(24):6481-6490. doi: 10.1182/bloodadvances.2025016701. PMID 40857358
- [Derived] Ligon JA, Cupit-Link MC, Yu C, Levine J, Foley T, Rotz S, Sharma A, Gomez-Lobo V, Shah NN. Pediatric Cancer Immunotherapy and Potential for Impact on Fertility: A Need for Evidence-Based Guidance. Transplant Cell Ther. 2024 Aug;30(8):737-749. doi: 10.1016/j.jtct.2024.06.006. Epub 2024 Jun 10. PMID 38866240
- [Derived] Frangoul H, Locatelli F, Sharma A, Bhatia M, Mapara M, Molinari L, Wall D, Liem RI, Telfer P, Shah AJ, Cavazzana M, Corbacioglu S, Rondelli D, Meisel R, Dedeken L, Lobitz S, de Montalembert M, Steinberg MH, Walters MC, Eckrich MJ, Imren S, Bower L, Simard C, Zhou W, Xuan F, Morrow PK, Hobbs WE, Grupp SA; CLIMB SCD-121 Study Group. Exagamglogene Autotemcel for Severe Sickle Cell Disease. N Engl J Med. 2024 May 9;390(18):1649-1662. doi: 10.1056/NEJMoa2309676. Epub 2024 Apr 24. PMID 38661449
- [Derived] Sharma A, Young A, Carroll Y, Darji H, Li Y, Mandrell BN, Nelson MN, Owens CL, Irvine M, Caples M, Jerkins LP, Unguru Y, Hankins JS, Johnson LM. Gene therapy in sickle cell disease: Attitudes and informational needs of patients and caregivers. Pediatr Blood Cancer. 2023 Jun;70(6):e30319. doi: 10.1002/pbc.30319. Epub 2023 Mar 28. PMID 36975201
- [Derived] Persaud Y, Mandrell BN, Sharma A, Carroll Y, Irvine M, Olufadi Y, Kang G, Hijano DR, Rai P, Hankins JS, Johnson LM. Attitudes toward COVID-19 vaccine among pediatric patients with sickle cell disease and their caregivers. Pediatr Blood Cancer. 2023 May;70(5):e30274. doi: 10.1002/pbc.30274. Epub 2023 Mar 1. PMID 36860093
- [Derived] Bhoopalan SV, Yen JS, Levine RM, Sharma A. Editing human hematopoietic stem cells: advances and challenges. Cytotherapy. 2023 Mar;25(3):261-269. doi: 10.1016/j.jcyt.2022.08.003. Epub 2022 Sep 17. PMID 36123234
- [Derived] Brusson M, Miccio A. Genome editing approaches to beta-hemoglobinopathies. Prog Mol Biol Transl Sci. 2021;182:153-183. doi: 10.1016/bs.pmbts.2021.01.025. Epub 2021 Mar 1. PMID 34175041
- [Derived] Frangoul H, Altshuler D, Cappellini MD, Chen YS, Domm J, Eustace BK, Foell J, de la Fuente J, Grupp S, Handgretinger R, Ho TW, Kattamis A, Kernytsky A, Lekstrom-Himes J, Li AM, Locatelli F, Mapara MY, de Montalembert M, Rondelli D, Sharma A, Sheth S, Soni S, Steinberg MH, Wall D, Yen A, Corbacioglu S. CRISPR-Cas9 Gene Editing for Sickle Cell Disease and beta-Thalassemia. N Engl J Med. 2021 Jan 21;384(3):252-260. doi: 10.1056/NEJMoa2031054. Epub 2020 Dec 5. PMID 33283989
- [Derived] Modarai SR, Kanda S, Bloh K, Opdenaker LM, Kmiec EB. Precise and error-prone CRISPR-directed gene editing activity in human CD34+ cells varies widely among patient samples. Gene Ther. 2021 Feb;28(1-2):105-113. doi: 10.1038/s41434-020-00192-z. Epub 2020 Sep 1. PMID 32873924